CLINICAL TRIAL: NCT06189157
Title: An Open-label Phase I/IIa, Multicentre, Interventional Single-arm Trial of MB-CART19.1 in Patients With Refractory SLE
Brief Title: MB-CART19.1 in Refractory SLE
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Miltenyi Biomedicine GmbH (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: M-2022-398
Record Dates: First submitted 2023-11-22; First posted 2024-01-03 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: SLE - Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Dose Level 0 (Experimental): Phase I: DL 0: 0,1x10e6 MB-CART19.1 cells Dose finding algorithm will start at dose level 1, with dose level 0 as a rescue dose.
  Interventions: Biological: MB-CART19.1
- Dose Level 1 (Experimental): Phase I: DL 1: 0,5x10e6 MB-CART19.1 cells Patients will be treated in cohorts of 3. If no DLT is determined, the dose can be escalated.
  Interventions: Biological: MB-CART19.1
- Dose Level 2 (Experimental): Phase I: DL 2: 1,0x10e6 MB-CART19.1 cells At the highest dose level 3 additional patients will be treated.
  Interventions: Biological: MB-CART19.1
- Phase II - Recommended dose MB-CART19.1 (Experimental): Phase II will evaluate the efficacy and safety in patients treated with the recommended dose
  Interventions: Biological: MB-CART19.1

INTERVENTIONS:
Biological: MB-CART19.1 — MB-CART19.1 consists of autologous CD19 Chimeric Antigen Receptor (CAR) transduced CD4/CD8 enriched T cells
  Other Names: CD19-targeting CAR T cells; Anti-CD19 CAR T cells

SUMMARY:
This is a phase l/ll open-label, multicentre, interventional single-arm trial of MB-CART19.1 in patients with refractory SLE systemic lupus erythematosus. In the phase I part, a maximum of n=12 patients will be treated in a maximum of 3 dose levels.

In the phase IIa part, a maximum of n=17 will be treated (n=10 patients in a 1st stage + n=7 patients in a 2nd stage). This includes the patients from the phase I part treated on the recommended dose level.

DETAILED DESCRIPTION:
Patients will be treated in cohorts of 3. After each cohort, the Safety Monitoring Board (SMB) will meet to assess whether the next higher dose level can be opened.

The follow-up of the patients will be performed in 3 steps:

* Until day 28 after treatment, the patients will be followed up closely by monitoring vital functions and lab parameters for signs of AEs and DLTs. Blood samples for the determination of persistence and phenotype of infused CAR+ cells will be taken. B cell aplasia in peripheral blood will be determined together with other secondary and exploratory biomarkers, response will be assessed and AEs will be documented.
* In the second follow-up phase until 1 year, blood samples for the determination of persistence and phenotype of infused CAR+ cells will be taken, B cell aplasia will be determined, response will be assessed and AEs will be documented until end of week 12, afterwards serious AEs (SAE) and AEs of special interest (AESI) will be documented, serious adverse reactions (SAR)/AESI will be reported.
* All patients irrespective of the clinical response will be followed up then for 1 more year or until the patient is lost to follow-up or has died. After completion of this last follow-up phase, patients will be rolled over to a subsequent follow-up observation for up to further 13 years.

ELIGIBILITY:
Inclusion Criteria:

1. Patients at least 18 years of age.
2. Signed and dated informed consent before the conduct of any trial-specific procedure.
3. SLE fulfilling the 2019 ACR/EULAR classification criteria (refer to Appendix 8).
4. One BILAG A or two BILAG B despite treatment with at least two of the following treatment options: MMF, cyclophosphamide, rituximab belimumab, anifrolumab, methotrexate, azathioprine.
5. SLE with major organ involvement defined as either:

   1. Presence of active lupus nephritis according to the following criteria:

      * Histology proven class III or IV lupus nephritis according to ISN/RPS 2003 classification
      * Urine protein-to-creatinine ratio (UPCR) >1 in 24-hour urine collection
      * Glomerular filtration rate (eGFR) of ≥30 mL/min/1.73 m2
      * No history of kidney transplantation.
   2. Lupus with heart involvement (e.g., myocarditis, pericarditis, endocarditis) as measured by MRI or echocardiography/ultrasound.
   3. Lupus with pulmonary involvement (Lupus pleuritis, pulmonary arterial hypertension (PAH)) or lung disease defined as:

      * Forced Vital Capacity (FVC) ≥ 60 % OR
      * Forced Expiratory Volume (FEV1) ≥ 60 %,Total Lung Capacity (TLC) ≥ 60 %, DLCO (diffusion capacity) ≥ 60 % (according to ATS/ERS guidelines).
6. Absolute CD3+ T cell count ≥ 100/µl.
7. No childbearing potential or negative pregnancy test at screening and before chemotherapy in women with childbearing potential. Subjects must agree to use a contraceptive method from screening until 12 months after the administration of the IMP.
8. Fully vaccinated against SARS-CoV-2 according to the recommendations of RKI or confirmed SARS-CoV-2 infection within the last 6 months.

Exclusion Criteria:

1. Active clinically significant central nervous system (CNS) dysfunction (including but not limited to uncontrolled seizure disorders, cerebrovascular ischemia or hemorrhage, dementia, paralysis).
2. Uncontrolled diabetes mellitus.
3. Therapy induced lung disease and tuberculosis.
4. Forced Vital Capacity (FVC) < 60 %, FEV1 < 60 %, Total Lung Capacity (TLC) < 60 % and DLCO (diffusion capacity) < 60 %.
5. BILAG A or BILAG B for neuropsychiatric SLE.
6. History of a malignancy unless disease free for ≥ 5 years with the exception of basal or squamous cell skin cancer.
7. Cardiac function: Unstable coronary heart disease; left ventricular ejection fraction (LVEF) < 50 %; no active myocarditis.
8. Renal function: eGFR < 30 ml/min/1.73 m2.
9. Liver function: Severe hepatic insufficiency defined as a Child-Pugh score > 10(C) (Appendix 10).
10. Known history of infection with human immunodeficiency virus or active infection with hepatitis B (hepatitis B surface antigen positive).
11. Known history of infection with hepatitis C virus unless treated and confirmed to be polymerase chain reaction (PCR) negative.
12. Any active, uncontrolled bacterial, viral or fungal infection including SARS-CoV-2.
13. History of hematopoietic stem cell or solid organ transplantation.
14. Irreversible organ damage.
15. Medications:

    * Systemic corticosteroids >10 mg within 7 days prior to leukapheresis;
    * T cell targeting drugs (e.g., mycophenolate mofetil, calcineurin inhibitors) within 21 days prior to leukapheresis;
    * Prior treatment with anti-CD19 therapy;
    * Previous adoptive T cell therapy or any gene therapy including CAR T cell therapy;
    * Live vaccines within 30 days prior to leukapheresis;
    * Current cytotoxic drugs.
16. Hypersensitivity against any drug or its ingredients/impurities that is scheduled or likely to be given during trial participation, e.g., as part of the mandatory preparative chemotherapy or rescue medication/salvage therapies for treatment related toxicities.
17. Contraindication of trial related procedures as judged by the investigator.
18. Women of childbearing potential (WOCBP) who do not agree to use highly effective contraceptive measures (Pearl index < 1) or practice true sexual abstinence from any heterosexual intercourse (true abstinence is only acceptable if it is in line with the preferred and usual life style of the participant) or have a vasectomised partner as the sole sexual partner (the vasectomised partner must have received medical assessment of the surgical success) for at least 1 month before the study start, during the study and in the 12 months following the last dose of study treatment.

    A woman is considered a WOCBP, i.e. fertile, following menarche and until becoming post-menopausal unless permanently sterile. WOCBP who want to become pregnant after completing treatment should seek advice about oocyte cryoconservation prior to treatment because of possible irreversible infertility. WOCBP must refrain from egg donation throughout the study until 12 months after the last dose of study treatment.

    Highly effective methods of contraception include hormonal contraceptives associated with inhibition of ovulation (oral, intravaginal, transdermal, injectable, implantable) and intrauterine devices or systems (e.g. hormonal and non-hormonal) and bilateral tubal occlusion.

    Permanent sterilization methods include hysterectomy, bilateral salpingectomy and bilateral oophorectomy.

    A post-menopausal state is defined as no menses for 12 months without an alternative medical cause.
19. Men with non-pregnant WOCBP partners who do not agree to use highly effective contraceptive measures (Pearl index < 1, e.g. spermicide and condom or other highly effective contraceptive measures (Pearl index < 1) taken by their WOCBP partner) or practice true sexual abstinence from any heterosexual intercourse (true abstinence is only acceptable if it is in line with the preferred and usual life style of the participant.), unless they are surgically sterile (meaning at least 2 consecutive analyses following vasectomy demonstrate absence of sperms in the ejaculate), during the study and in the 12 months following the last dose of study treatment.

    Men should seek advice about sperm conservation prior to treatment because of possible irreversible infertility. Men must furthermore refrain from sperm donation throughout the study until 12 months after the last administration of study treatment.
20. Concurrent participation in any other interventional trial.
21. Inability to understand the procedures and risks associated with the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2024-08-12 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Phase I: Determination of the recommended dose for phase IIa out of 3 dose levels | Until day 28 after infusion of MB-CART19.1
  Based on a Bayesian Optimal Interval (BOIN) design with DLT after infusion of MB-CART19.1
Phase I: Safety and toxicity of MB-CART19.1 | 24 months
  Incidence of adverse event (AE), classified according to CTCAE version 5.0, and evaluation and classification of Cytokine Release Syndrome (CRS) and Immune Effector cell-associated Neurotoxicity Syndrome (ICANS)
Phase IIa: Proportion of patients in remission after infusion of MB-CART19.1 | Month 6
  Remission is evaluated by fulfillment of DORIS remission criteria of SLE

SECONDARY OUTCOMES:
Phase I and Phase IIa: Treatment response to MB-CART19.1 | Day 28, Week 12, Month 6, Month 12, Month 24
  Measured by DORIS, LLDAS, SLEDAI 2K, BILAG
Phase I and Phase IIa: Patient reported outcomes | Day 0, Day 28, Week 12, Month 6, Month 12, Month 24
  SF-36, FACIT-F, HAQ-DI
Phase I and Phase IIa: Cellular and humoral immunogenicity | Day 28, Week 12, Month 6, Month 12
  Incidence of cellular and humoral immunogenicity
Phase I and Phase IIa: B cell aplasia and immunoglobulin deficiency | Day 0, all visits after Day 7 inclusive until Month 24
  Occurrence and duration of B cell aplasia, immunoglobulin levels
Phase I and Phase IIa: Levels of immunology parameters | Screening, Lymphodepletion, Day 0, Day 14, Day 28, Week 8, Week 12, Month 6, Month 9, Month 12, Month 24
  Changes in the levels of SLE associated serum autoantibodies, C3/C4, lupus anticoagulant
Phase I and Phase IIa: Persistence of MB-CART19.1 | All visits after Day 2 inclusive until Month 24
  Percentage of MB-CART19.1 of all T cells as well as total number of MB-CART19.1 in peripheral blood
Phase I and Phase IIa: Immunophenotyping of circulating immune cells | All visits starting from Day 0 inclusive
  Percentage of circulating immune cells and B-cell subsets measured by flow cytometry
Phase I and Phase IIa: Serum cytokines and BAFF | Day 14, Day 28, Week 8, Week 12, Month 6, Month 12
  Cytokine levels in peripheral blood

CONTACTS AND LOCATIONS:
Overall Officials: Georg Schett, Prof. Dr., Principal Investigator — University Clinical Erlangen, Medical Clinic 3
Locations (3):
- Germany (3):
  - Universitätsklinikum Erlangen, Medizinische Klinik 3, Erlangen
  - Otto-von-Guericke-Universität Magdeburg, Magdeburg
  - Universitatsklinikum Tubingen - Medizinische Universitätsklinik Abt. II, Tübingen

IPD SHARING:
Plan to Share IPD: No